CLINICAL TRIAL: NCT03770611
Title: Effect of a Nutritional Supplement of Probiotics and/or Prebiotics vs Placebo on Serum Concentrations of Uremic Toxins and Inflammatory Cytokines in Automated Peritoneal Dialysis Patients.
Brief Title: Effect of Prebiotics and/or Probiotics on Uremic Toxins and Inflammation Markers in Peritoneal Dialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Unidad de Investigacion Medica en Enfermedades Renales (Other)
Collaborators: Centro Universitario de Tonalá (Other); Universidad de Colima (Other)
Responsible Party: Principal Investigator, Alfonso Martín Cueto Manzano, Head of the Biomedical Research Unit 02, Unidad de Investigacion Medica en Enfermedades Renales
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: UIMER003
Record Dates: First submitted 2018-05-31; First posted 2018-12-10 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: End Stage Renal Failure on Dialysis
Keywords: dialysis; uremic toxin; inflammation; prebiotics; probiotics
MeSH Terms: conditions — Inflammation | interventions — Probiotics; Prebiotics

STUDY DESIGN:
Intervention Model Description: Parallel assignment, patients in automated peritoneal dialysis will be randomly assigned to one of the four intervention groups: probiotic, prebiotic, symbiotic and placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patient Blinding: Patients in automated peritoneal dialysis will be blinded to the intervention they will receive. Evaluator Blinding: The principal investigator and the Doctorate program student will be blinded to the intervention that patients will receive (probiotic, prebiotic, symbiotic or placebo).
  Care providers will be blinded to the intervention groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Probiotic (Active Comparator): Subjects receiving probiotic supplementation: 2x108 CFU probiotic bacteria + prebiotic placebo per day during 3 months
  Interventions: Dietary Supplement: Probiotic
- Prebiotic (Active Comparator): Subjects receiving prebiotic supplementation: 20 g of prebiotic fiber + probiotic placebo per day during 3 months
  Interventions: Dietary Supplement: Prebiotic
- Symbiotic (Experimental): Subjects receiving probiotic and prebiotic supplementation: 2x108 CFU probiotic bacteria + 20 g of prebiotic fiber per day during 3 months
  Interventions: Dietary Supplement: Symbiotic
- Placebo (Placebo Comparator): Subjects receiving placebo of probiotic and prebiotic per day during 3 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — The probiotic supplement is composed of the following bacterial strains: Bacillus coagulans, Bacillus subtilis, Bifidobacterium (B) bifidum, B. breve, B. longum, Lactobacillus (L) acidophilus, L. brevis, L. casei, L. helveticus, L. Paracasei, L plantarum, L. rhamnosus, L. salivarus, Lactococcus lactis, Pediococcus acidilactici, Pediococcus parvulus, Weisella confusa, Weisella paramesenteroides
  Arms: Probiotic
Dietary Supplement: Prebiotic — The prebiotic fiber is Agave inulin
  Arms: Prebiotic
Dietary Supplement: Symbiotic — The supplement is a combination of the probiotic product + the prebiotic fiber
  Arms: Symbiotic
Dietary Supplement: Placebo — The supplement is a combination of probiotic placebo and prebiotic fiber placebo. Placebo will consist on maltodextrin for both cases.
  Arms: Placebo

SUMMARY:
End-stage renal disease (ESRD) is a world public health problem, with high morbidity and mortality. Cardiovascular disease is the main cause of mortality in ESRD; uremic toxin retention and inflammation are considered non-traditional risk factors, as they have an active role in atherosclerosis and vascular calcification pathogenesis in dialysis patients.

Uremic toxins may be generated by internal protein metabolism, however, some toxins that can't be efficiently eliminated by dialysis such as indoxyl sulphate and p-cresyl sulphate (protein bound toxins), are generated by the microbial metabolism in the large intestine by proteolytic bacteria, and may diffuse easily through the intestinal lumen, as a leaky gut characterizes kidney disease.

The gut has been recognized as a potential source of inflammation in ESRD patients; accumulation of nitrogen compounds, presence of gastrointestinal symptoms, dietary changes and multiple drugs and supplements use, stimulates microbiota alterations as bacterial overgrowth and translocation. These phenomena, may active the immune system, promoting local and systemic inflammation, which in turn has negative effects increasing endothelial dysfunction, muscle catabolism, insulin and erythropoietin resistance, and decreases appetite.

Some methods have been proposed to decrease inflammation and uremic toxin accumulation, as more efficient dialysis and anti-inflammatory drugs; however, some of them have limited efficacy and high cost. Nutritional treatments focused on modifying intestinal environment, as pre- and probiotics have promising effects by altering production and absorption of uremic toxins and decreasing inflammation; nevertheless, there is scarce information regarding its use and their role in ESRD, particularly in peritoneal dialysis, which is a widely used therapy in México. Furthermore, there is no clinical study comparing the effectiveness of prebiotics, probiotics, and symbiotics on serum concentrations of uremic toxins and inflammation in ESRD patients. It is possible that the administration of a nutritional supplement of probiotics and/or prebiotics decreases the serum concentrations of uremic toxins and inflammation markers in ESRD patients on automated peritoneal dialysis compared to placebo.

DETAILED DESCRIPTION:
Objective:

The aim of the present study is to evaluate and to compare the effect of a nutritional supplement of probiotics and/or prebiotics on serum concentrations of uremic toxins and inflammatory markers compared to placebo, in automated peritoneal dialysis patients.

Sample size:

For the sample size calculation a mean differences formula was used, with a 95% confidence level, a 80% sample power and accuracy of 0.05. As a reference, the study of Salmean YA, 2015 was considered; in this study, the administration of pea fiber + inulin during 12 weeks in chronic kidney disease patients, significantly decreased (p<0.05) serum concentrations of p-cresol (5.82 ± 1.72 mg/L) in comparison to placebo (7.25 ± 1.74 mg/L). After substituting formula values and adding 20% of possible losses during follow-up, the sample size is: 28 patients.

Additionally, sample size calculation was made considering other outcomes. In the study of Xie LN, 2015, the administration of high-fermentable soluble fiber in ESRD patients on hemodialysis during 6 weeks, significantly decreased (p<0.05) inflammation markers: C-reactive protein (CRP), tumour necrosis factor alpha (TNFa) and interleukin 6 (IL-6) (4.8 ± 4.5 pg/mL, 10.1 ± 1.4 pg/mL, 31.8 ± 5.3 mg/L, respectively) compared to control group (9.5 ± 5.6 pg/mL, 13.1 ± 2.4 pg/mL, 51.5 ± 14.6 mg/L). After substituting the formula, sample size was 19, 7, and 5 for CRP, TNFa and IL-6, respectively.

Thus, the highest value was finally used: 28 patients for intervention group.

Statistical analysis:

Quantitative variables will be shown as mean and standard deviation or median (25-75 percentiles) according to their parametric or non-parametric distribution; Qualitative variables will be shown as frequency and percentage. Intergroup comparisons will be performed with χ2 or Fisher test for qualitative variables and one-way ANOVA or Kruskal-Wallis test for quantitative variables as appropriate. For intra-group comparisons Mc Nemar test will be used for qualitative variables and paired T-test, Wilcoxon, repeated-measures or Friedman ANOVA for quantitative variables as appropriate. An intention to treat analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* >3 months on automated peritoneal dialysis treatment
* Signed informed consent

Exclusion Criteria:

* ESRD of inflammatory cause (lupus, vasculitis, collagenopathies)
* Intake of probiotics, prebiotics or fiber in the last 3 months
* Use of anti-inflammatory drugs or nutritional supplements (immunossuppresants, pentoxifylline, NSAIDs, omega-3)
* Treated with antibiotics or sevelamer
* Treated with research drugs or participants in any clinical trial
* Peritonitis or active infection 2 weeks prior the study
* Any medical condition affecting intestinal absorption (inflammatory bowel disease, short bowel syndrome, bariatric surgery) or severe dysmotility
* Severe malnutrition
* Previous kidney transplantation
* Serious diseases altering the fina outcomes of the study: decompensated heart failure, chronic liver disease, cancer, AIDS.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2019-01-07 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Change of uremic toxins from basal to 1 and 3 months | Baseline, 1 month and 3 months
  Measurement of serum concentrations of the uremic toxins p-cresyl sulphate (mg/dL) and indoxyl sulphate (mg/dL) by means of liquid chromatography.
Change of uremic toxins from basal to 1 and 3 months | Baseline, 1 month and 3 months
  Measurement of serum concentrations of endotoxin (EU/mL) by means of Limulus amebocyte lisate test.

SECONDARY OUTCOMES:
Change in gut microbiota composition from basal to 1 and 3 months | Baseline, 1 month and 3 months
  Determination of fecal bacterial composition by DNA extraction and pyrosequencing analysis.
Change in gastrointestinal symptoms from basal to 1 and 3 months | Baseline, 1 month and 3 months
  Measurement of appetite and frequency and severity of gastrointestinal symptoms (nausea, vomiting, bloating, diarrhea, constipation) by means of a gastrointestinal symptoms questionnaire.
Change of inflammatory cytokines from basal to 1 and 3 months | Baseline, 1 month and 3 months
  Measurement of serum concentrations of inflammatory cytokines Interleukin-6 (pg/mL), Interleukin-10 (pg/mL) and Tumor Necrosis Factor alpha (pg/mL) by means of ELISA.
Change of inflammatory cytokines from basal to 1 and 3 months | Baseline, 1 month and 3 months
  Measurement of serum concentrations of C-Reactive Protein (mg/L) by means of nephelometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Umae Hospital de Especialidades, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Duranton F, Cohen G, De Smet R, Rodriguez M, Jankowski J, Vanholder R, Argiles A; European Uremic Toxin Work Group. Normal and pathologic concentrations of uremic toxins. J Am Soc Nephrol. 2012 Jul;23(7):1258-70. doi: 10.1681/ASN.2011121175. Epub 2012 May 24. PMID 22626821
- [Background] Gryp T, Vanholder R, Vaneechoutte M, Glorieux G. p-Cresyl Sulfate. Toxins (Basel). 2017 Jan 29;9(2):52. doi: 10.3390/toxins9020052. PMID 28146081
- [Background] Ito S, Yoshida M. Protein-bound uremic toxins: new culprits of cardiovascular events in chronic kidney disease patients. Toxins (Basel). 2014 Feb 20;6(2):665-78. doi: 10.3390/toxins6020665. PMID 24561478
- [Background] Vaziri ND, Yuan J, Norris K. Role of urea in intestinal barrier dysfunction and disruption of epithelial tight junction in chronic kidney disease. Am J Nephrol. 2013;37(1):1-6. doi: 10.1159/000345969. Epub 2012 Dec 19. PMID 23258127
- [Background] Schepers E, Glorieux G, Vanholder R. The gut: the forgotten organ in uremia? Blood Purif. 2010;29(2):130-6. doi: 10.1159/000245639. Epub 2010 Jan 8. PMID 20093818
- [Background] Hauser AB, Stinghen AE, Goncalves SM, Bucharles S, Pecoits-Filho R. A gut feeling on endotoxemia: causes and consequences in chronic kidney disease. Nephron Clin Pract. 2011;118(2):c165-72; discussion c172. doi: 10.1159/000321438. Epub 2010 Dec 16. PMID 21160227
- [Background] Lin CJ, Wu V, Wu PC, Wu CJ. Meta-Analysis of the Associations of p-Cresyl Sulfate (PCS) and Indoxyl Sulfate (IS) with Cardiovascular Events and All-Cause Mortality in Patients with Chronic Renal Failure. PLoS One. 2015 Jul 14;10(7):e0132589. doi: 10.1371/journal.pone.0132589. eCollection 2015. PMID 26173073
- [Background] Soleimani A, Zarrati Mojarrad M, Bahmani F, Taghizadeh M, Ramezani M, Tajabadi-Ebrahimi M, Jafari P, Esmaillzadeh A, Asemi Z. Probiotic supplementation in diabetic hemodialysis patients has beneficial metabolic effects. Kidney Int. 2017 Feb;91(2):435-442. doi: 10.1016/j.kint.2016.09.040. Epub 2016 Dec 4. PMID 27927601
- [Background] Wang IK, Wu YY, Yang YF, Ting IW, Lin CC, Yen TH, Chen JH, Wang CH, Huang CC, Lin HC. The effect of probiotics on serum levels of cytokine and endotoxin in peritoneal dialysis patients: a randomised, double-blind, placebo-controlled trial. Benef Microbes. 2015;6(4):423-30. doi: 10.3920/BM2014.0088. Epub 2015 Feb 12. PMID 25609654
- [Background] Salmean YA, Segal MS, Palii SP, Dahl WJ. Fiber supplementation lowers plasma p-cresol in chronic kidney disease patients. J Ren Nutr. 2015 May;25(3):316-20. doi: 10.1053/j.jrn.2014.09.002. Epub 2014 Nov 5. PMID 25446837
- [Background] Xie LM, Ge YY, Huang X, Zhang YQ, Li JX. Effects of fermentable dietary fiber supplementation on oxidative and inflammatory status in hemodialysis patients. Int J Clin Exp Med. 2015 Jan 15;8(1):1363-9. eCollection 2015. PMID 25785138
- [Background] Poesen R, Evenepoel P, de Loor H, Delcour JA, Courtin CM, Kuypers D, Augustijns P, Verbeke K, Meijers B. The Influence of Prebiotic Arabinoxylan Oligosaccharides on Microbiota Derived Uremic Retention Solutes in Patients with Chronic Kidney Disease: A Randomized Controlled Trial. PLoS One. 2016 Apr 21;11(4):e0153893. doi: 10.1371/journal.pone.0153893. eCollection 2016. PMID 27100399
- [Background] Viramontes-Horner D, Marquez-Sandoval F, Martin-del-Campo F, Vizmanos-Lamotte B, Sandoval-Rodriguez A, Armendariz-Borunda J, Garcia-Bejarano H, Renoirte-Lopez K, Garcia-Garcia G. Effect of a symbiotic gel (Lactobacillus acidophilus + Bifidobacterium lactis + inulin) on presence and severity of gastrointestinal symptoms in hemodialysis patients. J Ren Nutr. 2015 May;25(3):284-91. doi: 10.1053/j.jrn.2014.09.008. Epub 2014 Nov 6. PMID 25455039
- [Background] Cruz-Mora J, Martinez-Hernandez NE, Martin del Campo-Lopez F, Viramontes-Horner D, Vizmanos-Lamotte B, Munoz-Valle JF, Garcia-Garcia G, Parra-Rojas I, Castro-Alarcon N. Effects of a symbiotic on gut microbiota in Mexican patients with end-stage renal disease. J Ren Nutr. 2014 Sep;24(5):330-5. doi: 10.1053/j.jrn.2014.05.006. Epub 2014 Jul 22. PMID 25066654
- [Background] Rossi M, Johnson DW, Morrison M, Pascoe EM, Coombes JS, Forbes JM, Szeto CC, McWhinney BC, Ungerer JP, Campbell KL. Synbiotics Easing Renal Failure by Improving Gut Microbiology (SYNERGY): A Randomized Trial. Clin J Am Soc Nephrol. 2016 Feb 5;11(2):223-31. doi: 10.2215/CJN.05240515. Epub 2016 Jan 15. PMID 26772193
- [Derived] Cooper TE, Khalid R, Chan S, Craig JC, Hawley CM, Howell M, Johnson DW, Jaure A, Teixeira-Pinto A, Wong G. Synbiotics, prebiotics and probiotics for people with chronic kidney disease. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD013631. doi: 10.1002/14651858.CD013631.pub2. PMID 37870148